CLINICAL TRIAL: NCT05501353
Title: Explore Biomarkers Associated With Prognosis of Recurrent and Metastatic CRC After Secondary Radical Surgery by Multi-omics Methods
Brief Title: Explore Biomarkers Associated With Prognosis of Recurrent and Metastatic CRC After Surgery by Multi-omics Methods
Status: Recruiting | Type: Observational
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Collaborators: Guangzhou Burning Rock Dx Co., Ltd. (Industry); Guangdong Living Environment Harmless Treatment Center Co., Ltd. (Unknown)
Responsible Party: Sponsor
Other Study IDs: 2022-0465
Record Dates: First submitted 2022-07-31; First posted 2022-08-15 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2022-07

CONDITIONS: Colorectal Cancer Metastatic
Keywords: Colorectal Cancer; Colorectal Cancer Metastatic; multi-omics method; biomarker
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — During the study, the investigators collect two blood samples (a total of 7 blood samples, 10ml/sample) and one tissue sample (two cancer tissues and one adjacent cancer tissue, 50mg/sample) of subject
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Group1: Patients with various types of metastatic colorectal cancer who had underwent the radical resection of colorectal cancer and were planning to undergo radical resection of metastasis
  Interventions: Other: no intervention

INTERVENTIONS:
Other: no intervention — This study is an observational study, which does not affect the routine diagnosis and treatment of patients and only requires the collection of biological samples at specific nodes

SUMMARY:
This project is the first application, which is applied as a single center project and applied according to the screening quantity. This project is a multi-omics approach to explore biomarkers associated with prognosis after secondary radical resection of recurrent and metastatic colorectal cancer.

Main research objectives: 1. To detect DNA mutation and methylation in tumor tissues by NGS detection technology (the methylation dimension should be detected in adjacent tissues at the same time), and to explore specific molecular markers related to prognosis; 2. Using NGS test technology of blood in patients with preoperative and postoperative blood ctDNA mutations and methylation double dimension testing, respectively, to explore the preoperative and postoperative ctDNA mutations and the correlation between methylation status and recurrence, including but not limited to predict patients with recurrence of sensitivity, specificity, positive predictive value, negative predictive value and recurrence warning time and other indicators.

Main contents: This study intends to include single site for the first time/organ metastasis after radical treatment and surgical indications again in patients with colorectal adenocarcinoma (including but not limited to spread to the liver, lung metastasis, peritoneal metastasis, lymph node metastasis and other organ metastasis), collected in patients with preoperative peripheral blood and tissue samples, tissue adjacent to carcinoma and postoperative peripheral blood, NGS detection technology was used to detect DNA and mutation in the relevant samples, combined with clinical treatment and prognosis information of patients, and then explore biomarkers for predicting recurrence risk.

ELIGIBILITY:
Inclusion Criteria:

1. Colorectal cancer patients with first recurrence and metastasis after previous radical resection
2. Single site/organ metastasis is indicative of reoperation
3. Adenocarcinoma diagnosed by histology or cytology
4. At the time of signing the informed consent, the applicant must be 18 years old or older
5. Life expectancy is at least 12 weeks
6. ECOG score 0~1

Exclusion Criteria:

1. Currently participating in the intervention study treatment, or receiving other drugs or study devices within 4 weeks before enrollment
2. Concurrent with other malignant tumors
3. The investigator determined that the patient had other serious diseases that might affect follow-up and short-term survival
4. Cardiac function NYHA class III or IV heart disease
5. The presence of definite peripheral nerve disease
6. There is definite hearing loss
7. Other researchers think it is not suitable for inclusion

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with various types of metastatic colorectal cancer who had underwent the radical resection of colorectal cancer and are planning to undergo radical resection of metastasis
Sampling Method: Non-Probability Sample
Enrollment: 125 (Estimated)
Dates: Start 2022-07-22 (Actual); Primary Completion 2027-09-01 (Estimated); Study Completion 2027-09-01 (Estimated)

PRIMARY OUTCOMES:
molecular markers related to prognosis | up to 24 months
  The investigator collect preoperative peripheral blood, surgical tissue samples, adjacent tissues and postoperative peripheral blood from patients. DNA and mutation detection were performed on relevant samples using NGS detection technology and combined with clinical treatment and prognosis information of patients to explore the biomarkers (e.g. CtDNA mutation and ctDNA methylation were combined for MRD detection) of recurrence risk prediction.
the correlation between ctDNA mutations with methylation status and recurrence | up to 24 months
  using NGS test technology of blood in patients with preoperative and postoperative blood ctDNA mutations and methylation double dimension testing, respectively, to explore the correlation between the preoperative and postoperative ctDNA mutations with methylation status and recurrence, including but not limited to predict relapse in patients with sensitivity, specificity, positive predictive value, negative predictive value and recurrence warning time and other indicators;

SECONDARY OUTCOMES:
Compare the difference of DNA with ctDNA in predicting postoperative recurrence through statistical method | up to 24 months
  To compare the difference in the performance of DNA mutation dimension alone and ctDNA detection (DNA mutation + methylation dual dimension) in predicting postoperative recurrence through statistical method

CONTACTS AND LOCATIONS:
Overall Officials: Lifeng Sun, Study Director — 2ndAffiliated Hospital, School of Medicine, Zhejiang University, China
Locations (1):
- the Second Affiliated Hospital, Zhejiang University School of Medicine, Hangzhou, Zhejiang, China